CLINICAL TRIAL: NCT07346352
Title: Investigation of the Effect of Treadmill Training With Thera-Band on Depression, Mobility, Balance, and Gait in Stroke Patients: A Randomized Controlled, Single Blinded Study
Brief Title: Treadmill Training With Thera-Band in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Korkem, Assistant Professor, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.08.6.YÖK.2.ÜS.0.05.0.06/2018
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stroke Patients
Keywords: stroke; rehabilitation; balance; mobility; depression; treadmill; Thera-Band
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group received conventional physical therapy and treadmill walking training three days per week for eight weeks. Conventional therapy consisted of lower extremity weight-bearing and isolated joint exercises, bridge exercises, neuromuscular facilitation techniques, trunk rotation during reaching activities, standing training, spasticity-reducing exercises in sitting and lying positions, and activities of daily living training. Treadmill training was performed for 30 minutes per session at the participant's preferred walking speed, following an individualized familiarization protocol.
  Interventions: Other: Conventional therapy; Other: treadmill training
- Experimental Group (Experimental): Participants in the experimental group received Thera-Band-assisted resistance walking during treadmill training in addition to the same conventional therapy and treadmill protocol as the control group. A green Thera-Band providing approximately 2 pounds of resistance at 25% elongation was used for all participants. The band was applied to support the lower extremity during the swing phase and to facilitate foot placement, dorsiflexion, and eversion through elastic resistance and tactile stimulation.
  Interventions: Other: Conventional therapy; Other: treadmill training; Other: Thera-band

INTERVENTIONS:
Other: Conventional therapy — Conventional therapy consisted of lower extremity weight-bearing and isolated joint exercises, bridge exercises, neuromuscular facilitation techniques, trunk rotation during reaching, standing training, spasticity-reducing exercises in sitting and lying positions, and activities of daily living training
Other: treadmill training — Participants in each group were exercised on a Cateye EC-t220 model treadmill (Kuwazu, Higashi sumiyoshi-Ku, OSAKA, JAPAN) 3 days a week for 30 minutes each for 8 weeks. Every gait trial was conducted at the patient's chosen pace. Prior to the initial treadmill experiment, respondents were instructed to walk on the treadmill at a low belt speed (0.4 km/h 1) and increase the belt speed by 0.2 km/h 1 every 10 seconds until they reached their chosen gait speed without assistance. After around 30 seconds of maintaining this pace, the subjects were asked to reassess, and if required, the gait speed was changed. Until the patient's preferred walking speed was established, this procedure was repeated. Additionally, this procedure acted as a treadmill gait familiarization period. This acclimatization period was prolonged if needed until the participant reported having a comfortable gait while using the treadmill.
Other: Thera-band — In the intervention group, strengthening during treadmill training was provided using a green Thera-Band applied bilaterally to the lower extremities. The green Thera-Band was selected for all participants to standardize resistance, as it provides a moderate resistance of approximately 2 pounds at 25% elongation. The Thera-Band was wrapped around the distal foot, extended along the posterior aspect of the lower leg, passed behind the knee and in front of the thigh, and crossed over the dorsal surface of the ankle. This application aimed to support the lower limb during the swing phase and facilitate effective foot placement. Additionally, tactile stimulation along the lateral border of the foot was intended to facilitate dorsiflexion and eversion during gait.
  Arms: Experimental Group

SUMMARY:
Background: The aim of our study was to investigate the effects of treadmill training with Thera-Band on depression, mobility, balance, and gait in stroke patients.

Methods: This single-blind randomized controlled trial included 40 patients with hemiparesis (53.57±4.3 years). After assessment, patients were randomly assigned in two groups as intervention (Treadmill training + Thera-Band) and controls (Treadmill training). Before the intervention, participants in both groups received 30 minutes of convansional therapy and 30 minute treadmill training three times a week for 8 weeks. Intervention group additionally received Thera Band on both lower extremities. Patients' mobility levels were assessed using the Rivermead Motor Assessment Index (RMD), balance using the Berg Balance Scale (BBS), lower extremity spasticity using the Modified Ashworth Scale (MAS), depression levels using the Back Depression Scale, and gait ability using the footprint method on powdered ground. Assessments were repeated before and after 8 weeks of treatment.

Key words: stroke, rehabilitation, balance, mobility, depression, treadmill, Thera-Band

ELIGIBILITY:
Inclusion Criteria:

1. being 18 years of age or older,
2. being diagnosed with stroke for the first time,
3. being able to walk 10 meters independently,
4. having lower extremity spasticity below 3 according to the modified Ashword scale (MAS),
5. being between stages 3-4 according to Brunnstrom,
6. having a score of 22 or above on the mini mental test

Exclusion Criteria:

1. high blood pressure, heart disease,
2. agnosia or visual impairment,
3. limitation of joint movement in the lower extremity on the hemiplegic side,
4. any botulinum toxin application or surgical operation in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Mobility | 8 week
  Assessed using the Rivermead Mobility Index (RMI). A tool for assessing mobility status, including fundamental mobility activities, is the Rivermead Mobility Index (RMI). One question is based on the test-giver's observations, while the other fourteen are answered by the patient's self-report. From turning in bed to running, the RMI evaluates a variety of activities. The total score is between 0-15. The higher the score, the higher the mobility level of the individual
Balance | 8 week
  Assessed using the Berg Balance Scale (BBS). BBS is used to evaluate postural control and predict the risk of falls. The validity and reliability of the BBS has been demonstrated in both acute and chronic stroke patients. The 14 items on the BBS are scored on a total of 56 points, with 0-4 points awarded according on the patient's performance on each item. Impaired balance is indicated by 0-20 points, adequate balance is indicated by 21-40 points, and good balance is indicated by 41-56 points.
Walking Ability (Gait Parameters) | 8 week
  Assessed using the Footprint Method on a 10-meter powdered walkway. With the footprint method, footprints were obtained by walking on a 10 m powdered floor at the speed of their choice. The steps in the middle 6 m area were analyzed by subtracting 2 m at the beginning and 2 m at the end. With this method, intact side stride length, hemiplegic side stride length, double stride length, gait tempo (steps/minute) were determined.

SECONDARY OUTCOMES:
Lower Extremity Spasticity | 8 week
  Assessed using the Modified Ashworth Scale (MAS). Spasticity was assessed using the Modified Ashworth Scale (MAS), a widely used clinical tool that measures resistance during passive soft-tissue stretching.
  The scale grades muscle tone from 0 (no increase in muscle tone) to 4 (rigid in flexion or extension), with higher scores indicating greater spasticity.
Depression | 8 week
  Assessed using the Beck Depression Inventory (BDI). The Beck Depression Scale assesses depression's cognitive, emotional, and physical manifestations. There are twenty-one symptom categories on this self-assessment scale. 63 is the highest possible score. The severity of the depression increases with the total score. A score of 0-9 indicates little depression symptoms, 10-16 mild symptoms, 17-29 moderate symptoms, and 30-63 severe symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Special education and rehabilitation center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No